CLINICAL TRIAL: NCT04422106
Title: Predictors of Intestinal Anastomosis Leakage, Application of New Predictors and New Scores
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MD.19.10.239 - 2019/10/08
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-05

CONDITIONS: Anastomotic Leak
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Predictors of intestinal anastomosis leakage, application of new predictors and new scores — Early detection of disruption and leakage of intestinal anastomotic sites whether small or large intestine by using biochemical markers as predictors and indicators of leakage with application of scoring scale to assess presence or absence of leakage.

SUMMARY:
Aim of the work This study aims at; Early detection of disruption and leakage of intestinal anastomotic sites whether small or large intestine by using biochemical markers as predictors and indicators of leakage with application of scoring scale to assess presence or absence of leakage.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with intestinal or colonic anastomosis either elective or emergent.

Exclusion Criteria:

* Patients with inflammatory bowel disease will be excluded because this could influence plasma levels of inflammatory biomarkers.
* patients using corticosteroids
* Patients unfit for anaesthesia, those having collagen diseases or hematological disorders.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2020-06-17 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Early detection and management of intestinal anastomotic leak | 6 months
  Early detection of disruption and leakage of intestinal anastomotic sites whether small or large intestine by using biochemical markers as predictors and indicators of leak(Intestinal fatty acid binding protein, Procalcitonin and CRP) with application of scoring scale(Dekker et al 2011) (Dulk et al ., 2013) to assess presence or absence of leakage.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt